CLINICAL TRIAL: NCT05117307
Title: Comparison of Transversalis Fascia Plane Block and Erector Spinae Plane Blocks in Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Omer Doymus, Medical Doctor, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFP vs ESP on C/S
Record Dates: First submitted 2021-11-04; First posted 2021-11-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pain; Postoperative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): Ultrasound-guided erector spinae plane block with 20 ml %0.25 bupivacaine, per side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Group TFP (Active Comparator): Ultrasound-guided Transversalis Fascia Plane Block block with 20 ml %0.25 bupivacaine, per side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Ultrasound-guided block with 20 ml %0.25 bupivacaine, per side

SUMMARY:
Cesarean section is one of the most common major surgical procedures performed worldwide,, Post-cesarean analgesia should provide adequate pain control while allowing the mother to remain active to meet the needs of the baby. Insufficient analgesia after cesarean section may be associated with acute postoperative pain, chronic pain, higher opioid consumption, delayed functional capacity, and postpartum depression. Techniques such as neuraxial techniques, oral and intravenous agents, wound infiltration, and behavioral therapy can be used in the treatment of post-cesarean pain pain. In addition, Transversus abdominis plane block (TAP), Quadratus Lumborum block (QLB), Erector Spina block (ESP), Transversalis Fascia plane block (TFP) are used safely under ultrasound guidance. In this study, it was aimed primarily to examine the effects of TFP and ESP blocks on pain scores, and secondarily to evaluate analgesic consumption.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-50 years
* Cesarean Section

Exclusion Criteria:

* Cesarean Section under general anesthesia
* emergency cases
* those with a body mass index greater than 35 kg/m2
* coagulopathy
* local infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Postoperative first 24 hours
  Opioid consumption postroperative period

SECONDARY OUTCOMES:
Visual Analog Pain Score | Postoperative first 24 hours
  Pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Regional Training and Research Hospital, Erzurum, Yakutiye, Turkey (Türkiye)